CLINICAL TRIAL: NCT06803693
Title: A Study to Evaluate the Efficacy and Safety of Genotype-guided Targeted Agents in Combination With POLA-RCHP VERSUS POLA-RCHP in Patients With Previously Untreated Diffuse Large B-cell Lymphoma
Brief Title: Efficacy and Safety of Pola-RCHP-X vs Pola-RCHP in Untreated DLBCL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, M.D, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GUIDANCE05
Record Dates: First submitted 2025-01-27; First posted 2025-01-31 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — polatuzumab vedotin; Rituximab; Cyclophosphamide; Doxorubicin; Prednisone; zanubrutinib; Lenalidomide; Decitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pola-RCHP-X (Experimental): Participants will receive polatuzumab vedotin 1.8 milligrams per kilogram (mg/kg) intravenously (IV) on Day2, rituximab 375 milligrams per square meter (mg/m²) IV on Day 1, cyclophosphamide 750 mg/m² IV on Day 2， doxorubicin 50 mg/m² IV on Day 2 and prednisone 100 milligrams per day (mg/day) orally (PO) on Days 2-6 of every 21-day cycle for the first cycle. For the remaining 5 cycles, they will receive Zanubrutinib 160 mg BID PO on days 1-21, or lenalidomide 25 mg/day PO on days 1-10, or decitabine 10 mg/m²/day IV on days -5 to -1 followed by standard Pola-RCHP of every 21-day cycle.
  Interventions: Drug: Polatuzumab vedotin; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Prednisone; Drug: Zanubrutinib; Drug: Lenalidomide; Drug: Decitabine
- Pola-RCHP (Active Comparator): Participants will receive polatuzumab vedotin 1.8 milligrams per kilogram (mg/kg) intravenously (IV) on Day2, rituximab 375 milligrams per square meter (mg/m²) IV on Day 1, cyclophosphamide 750 mg/m² IV on Day 2， doxorubicin 50 mg/m² IV on Day 2 and prednisone 100 milligrams per day (mg/day) orally (PO) on Days 2-6 of every 21-day cycle for 6 cycles.
  Interventions: Drug: Polatuzumab vedotin; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Prednisone

INTERVENTIONS:
Drug: Polatuzumab vedotin — Polatuzumab vedotin IV infusion will be administered as per the schedule specified in the respective arm.
Drug: Rituximab — Rituximab IV infusion will be administered as per the schedule specified in the respective arm.
Drug: Cyclophosphamide — Cyclophosphamide IV infusion will be administered as per the schedule specified in the respective arm.
Drug: Doxorubicin — Doxorubicin IV infusion will be administered as per the schedule specified in the respective arm.
Drug: Prednisone — Prednisone PO will be administered as per the schedule specified in the respective arm.
Drug: Zanubrutinib — Zanubrutinib PO will be administered as per the schedule specified in the respective arm.
  Arms: Pola-RCHP-X
Drug: Lenalidomide — Lenalidomide PO will be administered as per the schedule specified in the respective arm.
  Arms: Pola-RCHP-X
Drug: Decitabine — Decitabine IV infusion will be administered as per the schedule specified in the respective arm.
  Arms: Pola-RCHP-X

SUMMARY:
The purpose of this study is to compare the efficacy and safety of genotype-guided targeted agents in combination with polatuzumab vedotin plus rituximab, cyclophosphamide, doxorubicin, and prednisone (Pola RCHP-X) versus Pola RCHP in Chinese patients with previously untreated diffuse large B-cell lymphoma (DLBCL).

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Age 18-75 years at the time of signing Informed Consent Form and willingness to comply with study protocol procedures
* Previously untreated participants with CD20-positive DLBCL
* IPI score 2-5
* ECOG Performance Status of 0, 1, or 2
* After 1 cycle of Pola-R-CHP, ctDNA decreased by < 3.0 LFC
* Life expectancy ≥ 6 months
* Left ventricular ejection fraction (LVEF) ≥ 50% on cardiac multiple-gated acquisition (MUGA) scan or cardiac echocardiogram (ECHO)
* Adequate hematologic function (unless due to underlying disease, as established for example, by extensive bone marrow involvement or due to hypersplenism secondary to involvement of the spleen by DLBCL per the investigator for which blood product transfusions are permitted) defined as follows:

  * Hemoglobin ≥ 9.0 g/dL without packed RBC transfusion during 7 days before first treatment
  * ANC ≥ 1.0 x 10^9/L
  * PLT ≥ 75 x 10^9/L

Exclusion Criteria:

* Contraindication to any of the individual components of Pola-RCHP or Zanubrutinib/Lenalidomide/ Decitabine
* Prior solid organ transplantation or SCT
* Current diagnosis of the following: Follicular lymphoma grade 3B; mediastinal grey zone lymphoma; primary mediastinal (thymic) large B-cell lymphoma; Burkitt lymphoma; PCNSL
* Significant or extensive history of cardiovascular disease such as New York Heart Association Class III or IV cardiac disease or Objective Assessment Class C or D, myocardial infarction within the last 6 months prior to the start of Cycle 1, unstable arrhythmias, or unstable angina
* History or presence of an abnormal ECG that is clinically significant in the investigator's opinion
* Any of the following abnormal laboratory values (unless any of these abnormalities are due to underlying lymphoma):

  * Serum AST and ALT ≥ 2.5 x ULN
  * Total bilirubin ≥ 1.5 x ULN
  * Serum creatinine clearance < 30 mL/min (using Cockcroft-Gault formula)
* Any active infection within 7 days prior to Cycle 1 Day 1 that would impact participant safety
* Positive test results for chronic hepatitis B infection (defined as positive hepatitis B surface antigen [HBsAg] serology)：Participants with occult or prior hepatitis B infection (defined as positive total hepatitis B core antibody and negative HbsAg) may be included if hepatitis B virus (HBV) DNA is undetectable at the time of screening. Such participants must be willing to undergo HBV DNA testing every month and appropriate antiviral therapy as indicated
* Positive test results for hepatitis C (hepatitis C virus [HCV] antibody serology testing)：Participants positive for HCV antibody are eligible only if PCR is negative for HCV RNA
* Participants with a history of progressive multifocal leukoencephalopathy
* Pregnancy or breastfeeding, or intention of becoming pregnant during the study or within 12 months after final dose of Pola-RCHP-X
* Other concurrent and uncontrolled medical conditions that, in the opinion of the investigator, would affect the patient's participation in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival（by IRC） | From randomization to the first occurrence of disease progression or relapse, or death from any cause, whichever occurs earlier (up to 24 months)
  PFS, defined as the time from randomization to the first occurrence of disease progression or relapse using the 2014 Lugano Response Criteria or death due to any cause, whichever occurs first; as determined by the investigator

SECONDARY OUTCOMES:
Progression-free survival（by the investigator） | From randomization to the first occurrence of disease progression or relapse, or death from any cause, whichever occurs earlier (up to 24 months)
  PFS, defined as the time from randomization to the first occurrence of disease progression or relapse using the 2014 Lugano Response Criteria or death due to any cause, whichever occurs first; as determined by the investigator
Event-free survival | up to approximately 24 months
  defined as the time from date of randomization to the earliest occurrence of any of the following:
  Disease progression/relapse as determined by the investigator and IRC (separately) Death due to any cause The primary efficacy reason determined by the investigator, other than disease progression/relapse, that leads to initiation of NALT If biopsy is obtained after treatment completion and is positive for residual disease regardless of whether NALT is initiated or not
Complete response rate | End of treatment visit (6-8 weeks after last dose on Day 1 of Cycle 6 [Cycle length=21 days]
  CR rate at the end of treatment by FDG-PET defined as the proportion of participants with CR at the end of treatment according to the 2014 Lugano Response Criteria; as determined by the investigator and IRC (separately)
Objective response rate | End of treatment visit (6-8 weeks after last dose on Day 1 of Cycle 6 [Cycle length=21 days]
  ORR at treatment completion or discontinuation defined as the proportion of participants with partial response (PR) or CR at the end of treatment according to the 2014 Lugano Response Criteria; as determined by the investigator and IRC(separately)
Overall survival | up to approximately 3 years
  OS defined as the time from randomization to death from any cause
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v5.0 | From enrollment to study completion, a maximum of 3 years
  An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai JiaoTong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No